CLINICAL TRIAL: NCT00441610
Title: An Extension Trial to a Phase I Dose Escalation Study of LBQ707 (Gimatecan) Administered Orally 5 Consecutive Days to Japanese Patients With Advanced Solid Tumor
Brief Title: An Extension Trial to a Phase I Dose Escalation Study of Gimatecan Administered Orally 5 Consecutive Days to Japanese Patients With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBQ707A1101E1
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-04

CONDITIONS: Advanced Solid Tumors
Keywords: Gimatecan; topoisomerase I inhibitor; advanced solid tumors
MeSH Terms: interventions — ST 1481

ARMS (1):
- Gimatecan (Experimental)
  Interventions: Drug: Gimatecan

INTERVENTIONS:
Drug: Gimatecan
  Other Names: LBQ707

SUMMARY:
CLBQ707A1101 assesses the tolerability, safety, efficacy and pharmacokinetics of gimatecan in Japanese patients.

ELIGIBILITY:
Inclusion criteria:

* Patients completing the core protocol (CLBQ707A1101, NCT00410358) exhibiting stable disease, or a partial or complete response as defined by the core protocol. If patients only have non-measurable lesions, he/she must not be exhibiting progressive disease

Exclusion criteria:

* Documented progressive disease as defined by the core protocol
* Patients with performance status of 3 or 4 on the ECOG scale

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by Adverse Events | 2.8 years
Anti-tumor activity assessed by RECIST criteria | 2.8 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Chiba, Japan

REFERENCES:
- See also: Results for CLBQ707A1101E1 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3946